CLINICAL TRIAL: NCT01444573
Title: Rate Ventricular Control Therapy by Implantable Continuous Monitor in Patients With Permanent Atrial Fibrillation
Brief Title: Rate Ventricular Control Therapy in Patients With Permanent Atrial Fibrillation
Acronym: REVEAL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RVL-001-32
Record Dates: First submitted 2011-09-29; First posted 2011-09-30 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Atrial Fibrillation
Keywords: Rate control; ILR
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 2 (Lenient control <120bpm) (Active Comparator)
  Interventions: Device: implantable continuous monitor
- Group 1 (Strict control <80 bpm) (Active Comparator)
  Interventions: Device: implantable continuous monitor

INTERVENTIONS:
Device: implantable continuous monitor — The Reveal XT was implanted in the parasternal area of the chest. The requirement for defining the exact final position was an R-wave amplitude ≥0.4 mV assessed through the Vector Check.
  Other Names: Reveal XT; implantable loop recorder

SUMMARY:
The investigators hypothesized that very lenient rate control is not inferior to strict or lenient rate control assessed by implantable continuous ECG monitor for preventing cardiovascular hospitalization and mortality in patients with long-standing persistent or permanent atrial fibrillation

ELIGIBILITY:
Inclusion Criteria:

* Long-standing persistent or permanent atrial fibrillation
* Mean resting heart rate > 80 beats per minute with or without rate control medication
* Age < 70 years old
* Constant use of anticoagulation therapy

Exclusion Criteria:

* Paroxysmal or persistent atrial fibrillation
* Non-stable heart failure or > III NYHA FC
* Indications for IPG/CRT/ICD
* Thyroid dysfunction
* Inability to walk or bike.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Hospitalization for all cardio-vascular events | 12 months

SECONDARY OUTCOMES:
All-cause death | 12 months
stroke | 12 months
life-threatening arrhythmic and drugs adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny A Pokushalov, MD, PhD, Principal Investigator — State Research Institute of Circulation Pathology
Locations (1):
- State Research Institute of CIrculation Pathology Novosibirsk, Russian Federation, Novosibirsk, Russia